CLINICAL TRIAL: NCT05070780
Title: Neurophysiological Evaluation of Muscle Tone in Healthy Subjects and in Patients With Increased Muscle Tone
Brief Title: Neurophysiological Evaluation of Muscle Tone
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Antonio Suppa, MD, PhD, Neuromed IRCCS
Other Study IDs: NEUR_02
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Muscle Tone Abnormalities; Rigidity, Muscle; Spasticity, Muscle
MeSH Terms: conditions — Muscle Rigidity; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Subjects
  Interventions: Device: Robot-assisted examination
- Patients with rigidity
  Interventions: Device: Robot-assisted examination
- Patients with spasticity
  Interventions: Device: Robot-assisted examination

INTERVENTIONS:
Device: Robot-assisted examination — evaluation of muscle tone with Robot-assisted perturbation

SUMMARY:
The primary objective of this study is to apply a biomechanical system (the NeuroFlexor) associated with the EMG recording to study the physiological mechanisms that contribute to the regulation of muscle tone in healthy subjects and in patients with increased muscle tone. A second fundamental objective of this study is to monitor over time the changes in muscle tone that can be found physiologically in healthy subjects and pathologically in patients with spasticy and/or rigidity. A further objective of this study is the quantitative evaluation of the symptomatic effects of specific therapies in improving the impaired muscle tone.

Clinical evaluation In this research project the investigators will recruit 20 patients with upper limb spasticity (regardless of the underlying disease responsible for the spasticity), 20 patients with Parkinson's disease characterized by stiffness of the upper limbs and 20 healthy control subjects. Patients will be recruited from the IRCCS Neuromed Institute, Pozzilli (IS). Participants will give their written informed consent to the study, which will be approved by the institutional ethics committee of the IRCCS Neuromed Institute, in accordance with the Declaration of Helsinki. All participants will be right-handed according to the Edinburgh handedness inventory (EDI) (Oldfield, 1971). Parkinson's disease will be diagnosed in accordance with the updated diagnostic criteria of the MDS (Postuma, RB et al. Validation of the MDS clinical diagnostic criteria for Parkinson's disease. Mov. Disord. Off. J. Mov. Disord. Soc. 33, 1601 -1608 (2018)., Nd). Clinical signs and symptoms of parkinsonian patients will be evaluated using the Hoehn & Yahr scale (H&Y), UPDRS part III (Patrick et al., 2001). The diagnosis of spasticity will be made through the neurological clinical evaluation of the patients and on the basis of the specific clinical history of the various pathologies underlying the spasticity itself (e.g. multiple sclerosis, stroke, spinal injuries). Spasticity will be assessed with the Modified Ashworth Scale "(MAS) (Harb and Kishner, 2021), the Modified Tardieu scale (MTS) (Patrick and Ada, 2006). Cognitive functions and mood, in both pathological conditions, will be evaluated using the clinical Mini-Mental State Evaluation (MMSE) scale (Folstein et al., 1975) and the Hamilton Depression Rating Scale (HAM_D) ( Hamilton, 1967). No participant must report pain problems and / or functional limitations affecting the upper limbs.

Exclusion criteria: - insufficient degree of passive wrist movement (<30 ° in flexion and <40 ° in extension) - tension at rest during NeuroFlexor recordings - hand pathologies (neurological or rheumatological) - upper limb fractures in the previous six months - presence of peacemakers or other stimulators - pregnancy.

All patients, and the group of healthy control subjects will have comparable anthropometric and demographic characteristics.

Experimental paradigm Participants will be seated comfortably, with the shoulder at 45 ° of abduction, the elbow at 90 ° in flexion, the forearm in pronation and the dominant hand placed on the platform of the Neuroflexor device. Participants will be instructed to relax during the test session, which will consist of the passive extension of the wrist at 7 speeds, one slow (5 ° / s) and 6 rapid (50 ° / s, 100 ° / s, 150 ° / s, 200 ° / s, 236 ° / s, 280 ° / s). The total range of wrist movement will be 50 °, starting from an initial angle of 20 ° in palmar flexion up to 30 ° in extension. Before the start of the experiment, participants will do practical tests in order to become familiar with the device. Two slow and five rapid movements will be made for each speed. The different angular velocities of wrist mobilization will be randomized. Slow movements will be performed before fast movements with an interval of 10 seconds between each test. For each participant, a NC, EC and VC value in Newton will be calculated by a dedicated software. The resistance profiles will also be obtained when the device was running idle (without hand) to allow the biomechanical model to isolate the forces originating from the hand from the intrinsic forces of the device. For each movement, the corresponding surface EMG trace will have been recorded, by placing the electrodes on the skin overlying the belly of the FRC and ERC muscles. An accelerometer, fixed on the back of the hand of the limb to be examined, will be used to synchronize the electromyograph with the NeuroFlexor. The EMG activity recorded by means of surface electrodes with belly-tendon type mounting, will be amplified using the Digitimer, will then be digitized at 5 kHz using the CED, and finally it will be stored on a computer dedicated to offline analysis. EMG recordings will be made at 6 speeds, 50°/ s, 100°/ s, 150°/ s, 200 °/s, 236 °/s, 280 °/s. For each trace the following parameters will be analyzed: latency, peak-to-peak amplitude and area of the EMG response.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* post-stroke spasticity

Exclusion Criteria:

* degenerative arthrosis
* rheumatoid arthritis
* cognitive impairment (MMSE <24)
* depression and other mood disorders (HAMD> 7)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy subjects, 20 Patients with rigidity, 20 Patients with spasticity, 20
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of biomechanical properties of muscles | 100 milliseconds
  total force

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Neuromed, Pozzilli, Italy

IPD SHARING:
Plan to Share IPD: Undecided